CLINICAL TRIAL: NCT04657250
Title: mHealth for Smoking Cessation in Public Housing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Lorien Abroms, PI, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCR191457
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Smoking Cessation
Keywords: mobile phone; mHealth; text messaging
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking cessation + quitline linkage text messages (Experimental): Text messaging for smoking cessation + text messages with proactive linkage to quitline
  Interventions: Behavioral: Smoking cessation + quitline linkage text messages
- Passive quitline referral (Placebo Comparator): Single text message with contact information for the Quitline
  Interventions: Behavioral: Passive quitline referral

INTERVENTIONS:
Behavioral: Smoking cessation + quitline linkage text messages — Smoking cessation text messages will provide behavioral skills and support for quitting smoking. Quitline linkage text messages will include contact information for the quitline, option to be contacted by the quitline and active referral to the quitline upon setting a Quit Date.
  Arms: Smoking cessation + quitline linkage text messages
Behavioral: Passive quitline referral — Single text message with contact information for the Quitline
  Arms: Passive quitline referral

SUMMARY:
Smoking rates among public housing residents are more than twice as high as in the general population. In August 2018, the U.S. Department of Housing and Urban Development (HUD) required all public housing in the U.S. to become smoke-free. While HUD recommended that Public Housing Authorities provide smoking cessations services, at present, the D.C. Housing Authority (DCHA) does not offer any cessation services to its residents. Low-income smokers face unique challenges to smoking cessation and require sustained support for smoking cessation. Digital interventions such as text messaging programs and quitline (QL) phone counseling are scalable, evidence-based interventions for smoking cessation that can provide support over an extended timeframe at low cost.

The aim of this proposed research is to conduct a feasibility trial to assess the acceptability, levels of engagement, and preliminary efficacy of an integrated program that combines text-messaging for smoking cessation and text messages providing proactive linkage to the quitline compared to a single passive quitline text message referral among DCHA residents. The investigators hypothesize that the integrated program (combining text messages for smoking cessation and proactive quitline linkage) will yield significantly higher rates of quit attempts than passive quitline referral only.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* resident of D.C. public housing
* smoked a cigarette in the 7 days prior to screening (self-report)
* has daily access to a working cell phone with an unlimited text message plan

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants making a quit attempt | 3 months
  not smoking for 24 hours or more because trying to quit smoking

SECONDARY OUTCOMES:
Proportion of participants who quit smoking | 3 months
  self reported 7 day point prevalence abstinence
Number of cigarettes smoked per day | 3 months
  change in number of cigarettes smoked per day between baseline and follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States